CLINICAL TRIAL: NCT05243810
Title: EPC Silver Wound Gel (EPC-123) Feasibility Clinical Study: Prospective, Single-arm, Repeated Measures Study of EPC Silver Wound Gel in the Management of Locally Infected Diabetic Foot Ulcers
Brief Title: EPC Silver Wound Gel (EPC-123) Feasibility Study in the Management of Mildly Infected Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Exciton Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-0279
Record Dates: First submitted 2022-01-11; First posted 2022-02-17 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Foot Ulcer; Non-healing Diabetic Foot Ulcer; Diabetic Foot Infection
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: A prospective, single-arm, repeated measures study feasibility study will be coordinated by the Lawson Health Research Institute on the use of EPC Silver Wound Gel (EPC-123) in patients with diabetic foot ulcers and localized infections within an outpatient clinical setting, to determine the safety of EPC Silver Wound Gel on diabetic foot ulcerations and impact on wound infection, wound ecology, and immunological biomarkers, in conjunction with the standard of care, to clarify parameters for a potential future study.
Masking Description: Patients will be assigned an internal ID number
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): A prospective, single-arm, repeated measures feasibility study will be coordinated on the use of EPC Silver Wound Gel in patients with diabetic foot ulcers and localized infections within an outpatient clinical setting, to determine the safety of EPC Silver Wound Gel on diabetic foot ulcerations and impact on wound infection classification, wound ecology, and immunological biomarkers, in conjunction with the standard of care, to clarify parameters for a potential future study.
  Interventions: Device: EPC Silver Wound Gel

INTERVENTIONS:
Device: EPC Silver Wound Gel — Re-application of EPC-123 will occur within 48 hours of the initial application. Secondary dressings will be selected at the discretion of the clinician or home care provider, based upon best practice guidelines for moisture management and will consist of a selection between the following secondary dressings: Mesorb® (Molnyke), Gauze, Cling (self-adherent gauze), or MediporeTM (3M). Application of EPC-123 will be executed at the Lawson Health Research Institute every second visit, where interim applications will be facilitated by home care. To support home care applications, a study kit will be provided to home care professionals inclusive of the EPC Silver Wound Gel, secondary dressings required, and instructions for removal/re-application.

SUMMARY:
The objective of this single-arm feasibility study is to investigate the safety and impact of the topical EPC Silver Wound Gel (EPC-123) in the management of diabetic foot ulcer wounds not progressing under the current standard of care.

DETAILED DESCRIPTION:
The objective of the proposed work is 1) to monitor clinical safety of EPC Silver Wound Gel on diabetic foot ulcers, 2) to evaluate the clinical impact of EPC Silver Wound Gel in foot ulcer progression in conjunction with the standard of care 3) to quantify the changes within the wound bacterial environment as it impacts wound healing and 4) to evaluate subjective patient and clinician outcomes: satisfaction, quality of life, perceived benefit, and compliance.

Consenting subjects who qualify for enrollment will proceed with two, weekly, visits related to screening. If screen passed, ie. under the current standard of care no progression of the diabetic foot ulcer is observed in accordance with validated diabetic foot ulcer classification metrics, then the subject will proceed with two weeks of study period where twice weekly clinic and twice weekly intermediate home-based care. This may be followed by an additional two weeks of study period, if warranted in accordance with best practice, with once weekly clinic and intermediate home care visits. In total there will be up to 9 clinic visits (minimum 7 clinic visits up to 9 clinic visits) in 6 weeks (screening and trial visits; minimum 4 weeks up to a maximum of 6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetes mellitus according to definitions outlined by the American Diabetes Association
* Presenting with an active or current foot ulcer that has been identified as stalled or persistent non-healing under current standard-of-care; showing no progression in 2 weeks as per IDSA guidelines.
* Presenting with a localized mild or local infection of the ulcer as listed in the IWGDF/IDSA Clinical Practice Guideline for the Diagnosis and Treatment of Diabetic Foot Infections (Table 1); exceeding 0.5 cm2 in area after appropriate debridement.
* Subject must agree to adhere to all protocol procedures and must be willing and able to provide written informed consent.
* Correction or optimization of underlying medical problems (e.g. diabetes or systemic infection).

Exclusion Criteria:

* Participants exhibiting extensive gangrene, and/or immediately limb-threatening infection
* Indications of osteomyelitis identified by plain radiographs taken within 2 days prior to study entry.
* No palpable dorsalis pedis or posterior tibial pulse or a pedal systolic pressure (Doppler ultrasound) of ≤ 40 mm Hg
* Clinically significant peripheral arterial disease requiring vascular intervention
* Patients requiring renal dialysis, immunosuppressive mediation, or those with uncontrolled hypertension.
* Lymphangitis; spread beneath the fascia; muscle, joint, or bone involvement.
* IDSA-defined severe infection, including systemic toxicity or metabolic instability
* Current use of enzymatic debridement.
* Participants with known silver sensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Incidence of intervention-related adverse events collected throughout the trial | Up to 28 days
  Clinical and/or biological adverse events will be reported over the intervention period. Severity of any adverse events will be graded.

SECONDARY OUTCOMES:
Qualitative improvement in quality of life assessment during the intervention period compared with screening period under standard of care. | Up to 28 days
  Quality of life will be assessed using the qualitative "Wound QoL" tool during the intervention period compared with qualitative assessment at baseline.
Progression of the Infectious Diseases Society of America and International Working Group on the Diabetic Foot Classifications of Diabetic Foot Infection during the intervention period compared with screening period under standard of care. | Up to 42 days
  Progressions of PEDIS (grade 1 = no symptoms or signs of infection; to grade 4, local infection with the signs of systemic inflammatory response syndrome) or IDSA Infection Severity (Uninfected; to Severe) during the intervention period compared with screening period under standard of care.
Progression the Diabetic Foot Infection (DFI) Wound Score during the intervention period compared with screening period under standard of care. | Up to 42 days
  Signs and symptoms of infection will be assessed using the 10-item DFI Wound Score system inclusive of semi-quantitative measurement of purulent discharge, non-purulent discharge, erythema, induration, tenderness, pain, warmth, size, depth, undermining. The DFI Wound Score ranges from a score of 3 (less severe wound) to 49 (more severe wound). Rate of change in DFI score during the intervention period will be compared with screening period under standard of care.
Progression the Bioburden Assessment Tool (BAT) during the intervention period compared with screening period under standard of care. | Up to 42 days
  The degree of bioburden will be assessed using BAT; measuring for the presence or absence of signs and symptoms of infection and bioburden and subsequent clinical interpretation. Progressions of the level of bioburden risk, from Category I (colonized: at risk) to Category VI (systemic infection), during the intervention period will be compared with screening period under standard of care.
Early clinical response | Within 48-72 hours of first intervention application
  Quantitation of lesion erythema area and wound area at 48-72 hours following the first intervention application.
Number of participants with systemic antibiotic or antifungal drug administration over the course of the intervention versus screening and baseline. | Up to 42 days
  Report on the number of participants receiving administration of systemic antibiotic or antifungal drugs during the intervention period compared with screening period under standard of care.
Progression in the absolute number of critical or qualified pathogen species present within the wound microbiome over the course of the intervention versus screening and baseline. | Up to 42 days
  Progression in the absolute number of critical or qualified pathogens (inclusive of those pathogens identified by the Centre for Disease Control and Prevention, World Health Organization, and the FDA as per 79 FR 32464) as per gene pyrosequencing over the course of intervention versus screening and baseline.
Progression in the relative quantity of critical or qualified pathogens versus commensal organisms present within the wound microbiome over the course of the intervention versus screening and baseline. | Up to 42 days
  Progression in the relative composition of critical or qualified pathogens (inclusive of those pathogens identified by the Centre for Disease Control and Prevention, World Health Organization, and the FDA as per 79 FR 32464) versus commensal organisms in the wound microbiome of as per gene pyrosequencing over the course of intervention versus screening and baseline.
Progression in wound microbiome over the course of the intervention versus screening and baseline. | Up to 42 days
  Progression of the wound microbiome on a whole ecology basis as per gene pyrosequencing; evaluating for community membership, structure, and diversity over the course of intervention versus screening and baseline.
Percent change in wound area and volume during the intervention period compared to baseline. | Up to 28 days
  Percent change in wound volume (cm3) at each visit compared to baseline.
Rate of wound closure, specifically percent change in area, during the intervention period compared with screening period under standard of care. | Up to 42 days
  Rate of wound closure, change in wound area (cm2), over the course of the intervention period compared to the screening period.
Rate of wound closure, specifically percent change in volume, during the intervention period compared with screening period under standard of care. | Up to 42 days
  Rate of wound closure, change in wound volume (cm3), over the course of the intervention period compared to the screening period.
Qualitative evaluation of patient satisfaction via questionnaire. | Up to 28 days
  Patient satisfaction over the course of the intervention period will evaluated. Patient satisfaction of the performance of the intervention will be evaluated within a rating scale of "poor" through to "excellent".
Qualitative evaluation of clinician satisfaction via questionnaire. | Up to 28 days
  Clinician satisfaction over the course of the intervention period will evaluated. Clinician satisfaction of the performance of the intervention will be evaluated within a rating scale of "poor" through to "excellent".
Progression of systemic biomarker C-Reactive protein (CRP). | Up to 28 days
  Quantitation of clinical change in CRP (mg/L) from baseline to end of intervention period.
Progression of systemic biomarker Erythrocyte sedimentation rate (ESR). | Up to 28 days
  Quantitation of clinical change in ESR (mm/hr) from baseline to end of intervention period.
Progression of systemic biomarker CBC and Differential. | Up to 28 days
  Quantitation of clinical change in CBC and Differential (cells per cubic millimeter) from baseline to end of intervention period.
Progression of systemic biomarker body temperature. | Up to 42 days
  Quantitation of clinical change in body temperature (degree Celsius) over the course of the intervention versus screening and baseline.
Progression in peri-wound microbiome over the course of the intervention versus screening and baseline. | Up to 42 days
  Progression of the peri-wound microbiome on a whole ecology basis as per gene pyrosequencing; evaluating for community membership, structure, and diversity over the course of intervention versus screening and baseline.
Quantitative progression of local inflammatory biomarkers over the course of the intervention versus screening and baseline. | Up to 42 days
  Quantitation of host inflammatory cytokines and chemokines (pg/ml) inclusive of: IL-1, IL-6, IL-8, IL-10 TNF-α, MMP-8, MMP-9, MMP-2, TIMP1, and TIMP2; within the wound over the course of the intervention versus screening and baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong DG, Swerdlow MA, Armstrong AA, Conte MS, Padula WV, Bus SA. Five year mortality and direct costs of care for people with diabetic foot complications are comparable to cancer. J Foot Ankle Res. 2020 Mar 24;13(1):16. doi: 10.1186/s13047-020-00383-2. PMID 32209136
- [Background] Boulton AJM, Armstrong DG, Hardman MJ, Malone M, Embil JM, Attinger CE, Lipsky BA, Aragon-Sanchez J, Li HK, Schultz G, Kirsner RS. Diagnosis and Management of Diabetic Foot Infections. Arlington (VA): American Diabetes Association; 2020 Jan. Available from http://www.ncbi.nlm.nih.gov/books/NBK554227/ PMID 32105420
- [Background] Lipsky BA, Berendt AR, Cornia PB, Pile JC, Peters EJ, Armstrong DG, Deery HG, Embil JM, Joseph WS, Karchmer AW, Pinzur MS, Senneville E; Infectious Diseases Society of America. 2012 Infectious Diseases Society of America clinical practice guideline for the diagnosis and treatment of diabetic foot infections. Clin Infect Dis. 2012 Jun;54(12):e132-73. doi: 10.1093/cid/cis346. PMID 22619242
- [Background] Lipsky BA, Polis AB, Lantz KC, Norquist JM, Abramson MA. The value of a wound score for diabetic foot infections in predicting treatment outcome: a prospective analysis from the SIDESTEP trial. Wound Repair Regen. 2009 Sep-Oct;17(5):671-7. doi: 10.1111/j.1524-475X.2009.00521.x. Epub 2009 Aug 11. PMID 19671126
- [Background] Lipsky BA, Senneville E, Abbas ZG, Aragon-Sanchez J, Diggle M, Embil JM, Kono S, Lavery LA, Malone M, van Asten SA, Urbancic-Rovan V, Peters EJG; International Working Group on the Diabetic Foot (IWGDF). Guidelines on the diagnosis and treatment of foot infection in persons with diabetes (IWGDF 2019 update). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3280. doi: 10.1002/dmrr.3280. PMID 32176444
- [Background] Blome C, Baade K, Debus ES, Price P, Augustin M. The "Wound-QoL": a short questionnaire measuring quality of life in patients with chronic wounds based on three established disease-specific instruments. Wound Repair Regen. 2014 Jul-Aug;22(4):504-14. doi: 10.1111/wrr.12193. PMID 24899053
- [Background] Houghton PE, Kincaid CB, Campbell KE, Woodbury MG, Keast DH. Photographic assessment of the appearance of chronic pressure and leg ulcers. Ostomy Wound Manage. 2000 Apr;46(4):20-6, 28-30. PMID 10788924